CLINICAL TRIAL: NCT02241083
Title: The Effect of Norepinephrine and Dopamine on Radial Forearm Free Flap Tissue Oxygen Pressure and Microdialysate Metabolite Measurements
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Minna Kääriäinen, MD, PhD, Senior Consultant, Associate Chief, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R05114
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Dopamine; Norepinephrine

ARMS (3):
- dopamine group (Active Comparator): vasopressor dosage individually titred according to the mean arterial pressure
  Interventions: Drug: Dopamine
- norepinephrine group (Active Comparator): vasopressor dosage individually titred according to the mean arterial pressure
  Interventions: Drug: Norepinephrine
- control group (Active Comparator): no medication
  Interventions: Other: no medication

INTERVENTIONS:
Drug: Dopamine
  Arms: dopamine group
Drug: Norepinephrine
  Arms: norepinephrine group
Other: no medication
  Arms: control group

SUMMARY:
Vasopressors may be needed after head and neck microvascular reconstructions to maintain sufficient mean arterial pressure. This is crucial for the flap survival. The study hypothesis is that norepinephrine and dopamine used as vasopressors do not affect flap tissue oxygen level and microdialysate metabolites.

ELIGIBILITY:
Inclusion Criteria:

* head and neck cancer patients having tumor ablation surgery and reconstruction with microvascular radial forearm flap

Exclusion Criteria:

* Patients having contraindications for the operation.
* Patient refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-06; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically definite ischemia in a flap confirmed by changes in tissue oxygen pressure level and microdialysates metabolites | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, P.O. Box 2000, Finland